CLINICAL TRIAL: NCT05221710
Title: Evaluation on the Effect of Acupuncture and Neuromuscular Electrical Stimulation on Mechanical Ventilation Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, JinyanXing, Director, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QYFYWZLL26719
Record Dates: First submitted 2022-01-09; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Insufficiency Requiring Mechanical Ventilation
Keywords: Respiratory Failure; weaning difficulty
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture Group (No Intervention): The acupuncture treatment will be performed by the technique of lifting, thrusting, twirling and rotating the needle until the patient is being "De-qi" (getting a numbness or other acupuncture feeling)
- Electroacupuncture Group (Experimental): On the basis of the above acupuncture treatment,two points that do not cross the joint will be chosen for electrical stimulation
  Interventions: Behavioral: electroacupuncture
- Neuromuscular Electrical Stimulation Group (No Intervention): Neuromuscular Electrical Stimulation(NMES) group received consecutive daily sessions of electrical stimulation at specific points

INTERVENTIONS:
Behavioral: electroacupuncture — The acupuncture treatment will be performed by the technique of lifting, thrusting, twirling and rotating the needle until the patient is being "De-qi" (getting a numbness or other acupuncture feeling).The needle will be kept in place for approximately 30 minutes. The point of acupuncture is determined by a traditional Chinese medicine doctor.
  Neuromuscular Electrical Stimulation(NMES) group received consecutive daily sessions of electrical stimulation at specific points.
  On the basis of the above acupuncture treatment,two points that do not cross the joint will be chosen for electrical stimulation in electroacupuncture group.
  Arms: Electroacupuncture Group

SUMMARY:
Acupuncture is a treatment intervention used globally for a wide variety of disorders. Its efficacy has been established over the course of 3000 years, originating in Asia and diversifying worldwide.The scientific basis for acupuncture remains unclear. Nonetheless, acupuncture releases neurochemical substrates, such as endorphins, serotonin, and norepinephrine.Acupuncture is considered to be a safe treatment when applied by a certified acupuncturist.Acupuncture has already been deployed in the treatment of sepsis or muscle weakness.Studies have revealed that acupuncture significantly improved grip strength and respiratory muscle strength in chronic obstructive pulmonary disease participates.Neuromuscular electrical stimulation (NMES) is an alternative to mobilize and exercise because it does not require active patient participation and can be used on bedridden patients.The investigators designed a study to compare the effects of acupuncture, electroacupuncture, and neuromuscular electrical stimulation on mechanical ventilation patients with weaning difficulties

ELIGIBILITY:
Inclusion Criteria:

* Prolonged mechanical ventilation duration (>72 h)
* stable oxygen saturation, fraction of inspired oxygen≤55%, and positive end expiratory pressure (PEEP)≤8 cmH2O
* dose of dopamine<10 μg/kg/min and dose of epinephrine<0.4 μg/kg/min;
* mean arterial pressure>75 mmHg and urine output>1 mL/kg/h
* good healing of the incision after surgery;
* normal cognitive function
* no history of chronic mental illness or chronic obstructive pulmonary disease

Exclusion Criteria:

* Inability to perform physical activities
* long-term MV prior to admission
* neurological comorbidities involving muscles
* irreversible disorders with a 6-month mortality rate of>50% according to Acute Physiology and Chronic Health Evaluation II (APACHEII)
* unsound limbs or unstable fractures
* administration of glucocorticoids (prednisone or other corticosteroid dose equivalents>20 mg/day) for at least 20 days prior to admission
* cardiopulmonary resuscitation before admission to the ICU
* radiotherapy or chemotherapy within the previous 6 months
* presence of comorbidities, including acute myocarditis, deep venous thrombosis/embolism, and cerebrovascular accident
* Patients with implanted pacemakers or defibrillators
* Pregnancy and lactation patients
* Patients with active bleeding or bleeding tendency
* Skin infection or injury at the acupuncture site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
ventilator-free days at 28 days | up to 28days

SECONDARY OUTCOMES:
Diaphragmatic thickening fraction(DTF) | baseline,Day 3 of mechanical ventilation,Day 7 of mechanical ventilation,before extubation
  DTF shows varied thickness of the diaphragm at end-expiration and end-inspiration. Te maximum and minimum values of each breathing cycle were taken as the end-inspiratory diaphragm thickness (DTei) and the end-expiratory diaphragm thickness (DTee), respectively. DTF was calculated by DTF=(DTei DTee)/DTee 100%. The values for 3 consecutive respiratory cycles were recorded and the average value was taken as the final value
Parasternal Intercostal Muscle Ultrasound | baseline,Day 3 of mechanical ventilation,Day 7 of mechanical ventilation,before extubation
  A 10-15 MHz linear array transducer was positioned perpendicular to the anterior thorax surface in the longitudinal scan, at the level of the second right intercostal space, approximately 6 to 8 cm lateral to the sternal edge with a window visualizing the second and third ribs. . Using M-mode, the ultrasound beam was perpendicularly directed at the midsection of the muscle, where it is the thinnest at end-expiration. The thickness of the parasternal intercostal muscle was measured on frozen images at end expiration and at peak inspiration.

CONTACTS AND LOCATIONS:
Overall Officials: Jinyan Xing, Dr., Study Director — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided